CLINICAL TRIAL: NCT03639467
Title: Phase Ib / II Study of Anlotinib Combined With Gemcitabine/Cisplatin in Previous Untreated Patients With Recurrent/Metastatic Nasopharyngeal Carcinoma
Brief Title: Study of Anlotinib Combined With Gemcitabine/Cisplatin in Advanced Nasopharyngeal Carcinoma
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Shi Yuankai, Vice President of Cancer Hospital Chinese Academy of Medical Sciences, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCC201807021
Record Dates: First submitted 2018-08-15; First posted 2018-08-21 (Actual); Last update posted 2018-09-18 (Actual); Status verified 2018-09

CONDITIONS: Recurrent Nasopharyngeal Carcinoma; Metastatic Nasopharyngeal Carcinoma
Keywords: anlotinib; nasopharyngeal carcinoma; gemcitabine; cisplatin
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — anlotinib; Gemcitabine; Cisplatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Anlotinib plus gemcitabine/cisplatin (Experimental): In the phase Ib portion, patients received dose escalation of anlotinb (from 8mg to 12mg orally once daily on days 1-14 of a 21-day) in combination with fixed dose of gemcitabine (1000mg/m2 intravenously on days 1 and 8) and cisplatin (80mg/m2 intravenously on day 1) every 3 weeks.
  In the phase II portion, patients received anlotinb at recommended phase II dose determined in the phase Ib portion, in combination with fixed dose of gemcitabine and cisplatin every 3 weeks.
  The combination of anlotinib plus gemcitabine / cisplatin was repeated every 3 weeks for up to six cycles. Patients with disease control (defined as a complete response, a partial response, or stable disease) continue to receive anlotinb until disease progression or unacceptable toxic effects, whichever occurred first.
  Interventions: Drug: Anlotinib plus gemcitabine/cisplatin

INTERVENTIONS:
Drug: Anlotinib plus gemcitabine/cisplatin — In the phase Ib portion, patients received dose escalation of anlotinb (from 8mg to 12mg orally once daily on days 1-14 of a 21-day) in combination with fixed dose of gemcitabine (1000mg/m2 intravenously on days 1 and 8) and cisplatin (80mg/m2 intravenously on day 1) every 3 weeks.
  In the phase II portion, patients received anlotinb at recommended phase II dose determined in the phase Ib portion, in combination with fixed dose of gemcitabine and cisplatin every 3 weeks.
  The combination of anlotinib plus gemcitabine / cisplatin was repeated every 3 weeks for up to six cycles. Patients with disease control (defined as a complete response, a partial response, or stable disease) continue to receive anlotinb until disease progression or unacceptable toxic effects, whichever occurred first.

SUMMARY:
Gemcitabine plus cisplatin (GC) is more effective than fluorouracil plus cisplatin in the treatment of recurrent or metastatic NPC (R/M-NPC). GC is the standard first-line chemotherapy regimen for this population. However, the median progression-free survival was only 7 months for GC regimen. Anlotinib is a kinase inhibitor of receptor tyrosine with multi-targets, especially for VEGFR2、VEGFR3、PDGFRβ and c-Kit, which has strong effect of anti-angiogenesis. This study is aim to evaluate the efficacy and safety of the combination regimen of anlotinib plus GC as first-line treatment for R/M-NPC.

DETAILED DESCRIPTION:
In the phase Ib portion, an escalated dose cohort is recruited to determine the maximum tolerated dose (MTD) and recommended phase II dose (RP2D) of anlotinib when given in combination with gemcitabine/cisplatin. The phase II portion is designed to characterize the efficacy and safety of the combination therapy in previous untreated patients with R/M-NPC.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years to 70 years.
2. Histological/cytological confirmation of NPC.
3. Primarily metastatic (stage IVB as defined by the International Union against Cancer and American Joint Committee on Cancer staging system for NPC, eighth edition) or recurrent NPC that is not amenable for local regional treatment or curative treatment.
4. Patients did not receive systemic chemotherapy for recurrent or metastatic disease, except for prior induction, concurrent, or adjuvant chemotherapy that was completed > 6 months prior to registration. Prior radiotherapy or chemoradiotherapy should be completed > 6 months prior to registration;
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0 - 1.
6. Life expectancy of more than 12 weeks.
7. At least one measurable lesion according to RECIST 1.1 which has not received radiotherapy ≥ 3 months.
8. Adequate hepatic, renal, heart, and hematologic functions: absolute neutrophil count (ANC) ≥ 1.5×109/L, platelet count (PLT) ≥ 100×109/L, hemoglobin (HB) ≥ 90 g/L, total bilirubin (TBIL) ≤ 1.5×upper limit of normal (ULN), alternate aminotransferase (ALT) or aspartate aminotransferase (AST) ≤ 3×ULN (or ≤ 5×ULN in patients with liver metastases), Serum Cr ≤ 1×ULN, Cr clearance ≥ 60 mL/min, international normalized ratio (INR) < 1.5 or prothrombin time (PT) < ULN+4s or activated partial thromboplastin time (APTT) < 1.5×ULN, proteinuria < (++) or urinary protein ≤ 1.0 g/24 hrs;
9. For women of child-bearing age, the pregnancy test results (serum or urine) within 7 days before enrolment must be negative. They will take appropriate methods for contraception during the study until the 8th week post the last administration of study drug. For men (previous surgical sterilization accepted), will take appropriate methods for contraception during the study until the 8th week post the last administration of study drug.
10. Signed informed consent.

Exclusion Criteria:

1. Other malignancy within the past five years other than basal cell skin cancer, or carcinoma in situ of the cervix;
2. Factors affecting the oral medication (e.g. inability to swallow, chronic diarrhea and intestinal obstruction);
3. Major injuries and/or surgery ≤ 4 weeks prior to registration with incomplete wound healing.
4. Patients with poor-controlled arterial hypertension (systolic pressure ≥ 140 mmHg and/or diastolic pressure ≥ 90 mm Hg) despite standard medical management;
5. Suffered from grade II or above myocardial ischemia or myocardial infarction, uncontrolled arrhythmias. Grade III-IV cardiac insufficiency according to New York Heart Association (NYHA) criteria or echocardiography check: left ventricular ejection fraction (LVEF)<50%;
6. History of clinically significant haemoptysis ≤ 2 months (more than half of one tea spoon of fresh blood per day) prior to registration. Coagulation disfunction, hemorrhagic tendency or receiving anticoagulant therapy;
7. History of clinically relevant major bleeding event (e.g. gastrointestinal hemorrhage, bleeding ulcer, occult blood ≥ (++), and vasculitis) ≤ 3 months prior to randomization;
8. Patients who have active brain metastases or leptomeningeal disease. Patients with treated brain metastases are eligible if they are clinically stable with regard to neurologic function, off steroids after cranial irradiation ending at least 3 weeks prior to randomization, or after surgical resection performed at least 3 weeks prior to randomization. No evidence of Grade greater than or equal to 1 central nervous system (CNS) hemorrhage based on pretreatment CT or MRI scan; Centrally located tumors of local invasion of major blood vessels, or distinct interstitial lung disease by the chest radiographic findings (CT or MRI);
9. Treatment with other investigational drugs or other anti-cancer therapy;
10. Previous therapy with anti-angiogenic drugs (such as anlotinib, apatinib, bevacizumab, endostar, etc.)
11. Treatment in another investigational trial ≤ 4 weeks prior to registration;
12. History of hypersensitivity to anlotinib, gemcitabine, cisplatin and/or the excipients of the trial drugs;
13. Active or chronic hepatitis C and/or B infection, or other active uncontrolled infection;
14. History of immunodeficiency disease (including HIV positive), concurrent acquired or congenital immunodeficiency syndrome, or history of organ transplantation;
15. History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess ≤ 6 months prior to registration;
16. History of arterial or venous thromboembolic events (e.g. cerebrovascular accident, cardiovascular accident, deep venous thrombosis and pulmonary embolism) ≤ 12 months prior to randomization;
17. Evidence of significant medical illness that in the investigator's judgment will substantially increase the risk associated with the subject's participation in and completion of the study;
18. History of mental diseases;
19. Other conditions regimented at investigators' discretion.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-09-18 (Estimated); Primary Completion 2021-08-22 (Estimated); Study Completion 2023-08-15 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | up to 3 years
  From date of enrollment until the date of first documented progression or date of death from any cause,whichever came first

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | up to 3 years
  The objective Response Rate of anlotinib plus gemcitabine/cisplatin in Previous Untreated Patients With Recurrent/Metastatic Nasopharyngeal Carcinoma
Overall survival (OS) | up to 3 years
  OS of of anlotinib plus gemcitabine/cisplatin in previous untreated patients with recurrent/metastatic Nasopharyngeal Carcinoma
Incidence of treatment-emergent adverse events (safety and tolerability) | up to 3 years
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.03

CONTACTS AND LOCATIONS:
Overall Officials: Yuankai Shi, MD, Principal Investigator — ChineseAMS
Locations (1):
- National Cancer Center/Cancer Hospitial,Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Han B, Li K, Zhao Y, Li B, Cheng Y, Zhou J, Lu Y, Shi Y, Wang Z, Jiang L, Luo Y, Zhang Y, Huang C, Li Q, Wu G. Anlotinib as a third-line therapy in patients with refractory advanced non-small-cell lung cancer: a multicentre, randomised phase II trial (ALTER0302). Br J Cancer. 2018 Mar 6;118(5):654-661. doi: 10.1038/bjc.2017.478. Epub 2018 Feb 13. PMID 29438373